CLINICAL TRIAL: NCT02143388
Title: Concurrent Cisplatin Chemoradiation With or Without Capecitabine as Adjuvant Chemotherapy in Local Advanced High Risk Nasopharyngeal Carcinoma: Randomized Control Clinical Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhao Chong (Other)
Collaborators: Jiangxi Provincial Cancer Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor-Investigator, Zhao Chong, MD, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCRT-AC-LAHR-NPC
Record Dates: First submitted 2014-05-07; First posted 2014-05-21 (Estimated); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Local Advanced High Risk Nasopharyngeal Carcinoma
Keywords: Local advanced; high risk; nasopharyngeal carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiation + adjuvant chemotherapy (Experimental): IMRT combine with cisplatin concurrent chemotherapy plus capecitabine adjuvant chemotherapy
  Interventions: Drug: IMRT combine with cisplatin concurrent chemotherapy plus capecitabine adjuvant chemotherapy
- Concurrent chemoradiation (Active Comparator): IMRT combine with cisplatin concurrent chemotherapy
  Interventions: Drug: IMRT combine with cisplatin concurrent chemotherapy

INTERVENTIONS:
Drug: IMRT combine with cisplatin concurrent chemotherapy — Patients in the control arm received radical radiotherapy with IMRT, and cisplatin (100mg/m2 on day 1) every three weeks for three cycles during RT.
  Arms: Concurrent chemoradiation
Drug: IMRT combine with cisplatin concurrent chemotherapy plus capecitabine adjuvant chemotherapy — Patients in the experimental arm received radical radiotherapy with IMRT, and cisplatin (100mg/m2 on day 1) every three weeks for three cycles during RT,followed by adjuvant chemotherapy with oral capecitabine(1000mg/m2/ twice a day for 14 days)every three weeks for eight cycles.
  Arms: Concurrent chemoradiation + adjuvant chemotherapy

SUMMARY:
This is an randomized controlled, multicenter clinical trial. The purpose of this study is to evaluate acute toxicity and efficacy of concurrent cisplatin chemoradiation with or without capecitabine as adjuvant chemotherapy in local advanced high risk nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Newly histologic diagnosis of nasopharyngeal carcinoma(WHO II/III)
* Clinical stage III~IVb(UICC 7th)
* Meet at least one factor below :1 primary tumor SUVmax>10 in 18F-FDG PET/CT;2 primary tumor volume>30cm3;3 mutiple metastatic cervical lymph node with at least one's short diameter>4cm; 4 T4N2M0; 5 T1-4N3M0;6 EBV-DNA>2×10E4 copy/l
* Range from 18～70 years old
* WBC count ≥ 4×109/L，Hemoglobin ≥ 100g/L， platelet count ≥ 100×109/L
* ALT or AST < 2.5×ULN、bilirubin < 1.5×ULN
* OSerum creatinine < 1.5×ULN

Exclusion Criteria:

* Central nervous system metastases
* Suitable for local treatment
* Uncontrolled seizure disorder or other serious neurologic disease
* Clinically significant cardiac or respiratory disease
* Drug or alcohol addition
* Do not have full capacity for civil acts
* Severe complication, active infection
* Concurrent immunotherapy or hormone therapy for other diseases
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Failure free survival | 3-year
  Defined as the time from date of recruitment to documented relapse or death from any cause.

SECONDARY OUTCOMES:
Acute Toxicity | 18 months
  To evaluate the acute toxicity with CTC 3.0 when concurrent cisplatin chemoradiation with or without capecitabine as adjuvant chemotherapy is used.

OTHER OUTCOMES:
Locoregional relapse free survival | 3-year
  Defined as the time from date of recruitment to documented locoregional relapse or death from any cause.
Distance metastasis free survival | 3-year
  Defined as the time from date of recruitment to documented distant metastatic recurrence or death from any cause.
Overall survival rate | 3-year
  Defined as the time from date of recruitment to death from any cause.
Late Toxicity | 3 years
  To evaluate the late toxicity with the RTOG/EORTC criterion when concurrent cisplatin chemoradiation with or without capecitabine as adjuvant chemotherapy is used.

CONTACTS AND LOCATIONS:
Overall Officials: zhao chong, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu Y, Yan W, Chen Y, Miao J, Zhang H, Wang J, Zhang Y, Huang X, Wang K, Qu Y, Chen X, Zhang J, Luo J, Li YX, Zhao C, Ma J, Wu R, Yi J. Treatment response-adapted risk index model for survival prediction and adjuvant chemotherapy selection in nonmetastatic nasopharyngeal carcinoma. NPJ Digit Med. 2025 Sep 1;8(1):564. doi: 10.1038/s41746-025-01918-2. PMID 40890288
- [Derived] Miao J, Wang L, Tan SH, Li JG, Yi J, Ong EHW, Tan LLY, Zhang Y, Gong X, Chen Q, Xiang YQ, Chen MY, Guo Y, Lv X, Xia WX, Tang L, Deng X, Guo X, Han F, Mai HQ, Chua MLK, Zhao C. Adjuvant Capecitabine Following Concurrent Chemoradiotherapy in Locoregionally Advanced Nasopharyngeal Carcinoma: A Randomized Clinical Trial. JAMA Oncol. 2022 Oct 13;8(12):1776-85. doi: 10.1001/jamaoncol.2022.4656. Online ahead of print. PMID 36227615
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn